CLINICAL TRIAL: NCT06260969
Title: Endovascular Treatment of Acute Ischemic Stroke With Underlying Intracranial Artery Stenosis: a Prospective, Multicentre Registry Study
Brief Title: Endovascular Treatment of Acute Ischemic Stroke With Underlying Intracranial Artery Stenosis
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Director, Head of Neurosurgery, Principal Investigator, Clinical Professor, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2023-WM13
Record Dates: First submitted 2023-12-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Large Vessel Occlusion; Intracranial Artery Occlusion With Cerebral Infarction; Endovascular Treatments; Acute Ischemic Stroke
Keywords: Endovascular treatments; Acute ischemic stroke; Stroke etiology; Retrieved clots; Intracranial artery stenosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — Thrombosis specimens；Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Endovascular therapy: Direct balloon dilation vs stenting vs embolectomy + tirofiban vs embolectomy + balloon dilation vs embolectomy + balloon dilation + intracranial stenting
  Interventions: Device: balloon dilatation

INTERVENTIONS:
Device: balloon dilatation — Direct balloon dilation vs stenting vs embolectomy + tirofiban vs embolectomy + balloon dilation vs embolectomy + balloon dilation + intracranial stenting
  Other Names: endovascular stenting; aspiration catheter; stent retriever; Tirofiban; intracranial stenting; normal saline

SUMMARY:
The study is a prospective multicentre registry study. Patients admitted to 10 stroke centres nationwide from September 2022 to September 2025 with acute ischaemic stroke due to large vessel occlusion considering underlying ICAS and treated with emergency endovascular thrombolysis were included for analysis. Patients who met the general inclusion criteria underwent thrombectomy and the necessary remedial treatment.

DETAILED DESCRIPTION:
The focus of this trial is to investigate the neuroprotective effects of endovascular hypothermia on the refractory disease of large vessel occlusion with underlying ICAS by performing different modes of endovascular interventions including stenting, balloon dilationand balloon dilation combined with stenting in patients who meet clinical and imaging criteria. The clinical prognosis of patients with different treatment modalities will be followed up to provide high quality clinical evidence to guide the interventional treatment of potential large vessel occlusions in ICAS. The main objectives of the study were to establish a prospective cohort of acute large vessel occlusions with potential ICAS treated with endovascular therapy based on the specific etiology of stroke with a high prevalence of intracranial atherosclerotic stenosis in the Chinese population; to explore the efficacy and safety of endovascular therapy for acute ischaemic stroke with potential ICAS; to investigate the use of different endovascular treatment modalities for acute ischaemic stroke with potential ICAS in the Chinese population; and to explore the neuroprotective effects of selective endovascular hypothermia on large vessel occlusions with potential ICAS. To explore the neuroprotective effect of selective endovascular hypothermia on large vessel occlusion in potential ICAS. To provide objective data and theoretical support for the choice of treatment for large vessel occlusion in underlying ICAS

ELIGIBILITY:
Inclusion Criteria:

* CT scan to exclude intracranial haemorrhage；CT angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography showing occlusion of the distal intracranial carotid artery or the first segment of the middle cerebral artery；ELVO with a base ICAS of > 70%；Mechanical thrombectomy within 6h after symptom onset in ischemic stroke；NIHSS≥6；receiving endovascular treatments；informed consent form signed by the patient or their legal representatives.

Exclusion Criteria:

* Hemorrhagic body, coagulation factor deficiency or oral anticoagulant therapy(INR > 3.0)；Baseline platelet count <50,000/µL；Baseline blood glucose <50mg/dL or >400mg/dL；Intractable hypertension(systolic blood pressure >220 mmHg or diastolic blood pressure >110 mmHg) that cannot be controlled by medication；Patients intubated without a NIHSS score assessed by a neurologist or emergency physician prior to intubation；Stroke attack with epilepsy affecting baseline NIHSS score；End-stage diseases leading to less than one year of expected survival for patients；Severe allergy to contrast media；Patients with renal insufficiency (blood creatinine ≥ 3 mg/dL)；Female patients who are pregnant or breastfeeding；The patient is participating in other drugs or device studies that may affect this study；Patient with cerebral vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral infarction with underlying intracranial artery stenosis receiving endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a clinical prognosis of mRS 0-2 at 90 days | patients achieve a clinical prognosis of mRS 0-2 at 90 days
  Proportion of patients achieving a clinical prognosis of mRS 0-2 at 90 days

SECONDARY OUTCOMES:
Proportion of patients with a good prognosis early after treatment | 24 hours after thrombectomy
  Decrease in NIHSS score ≥ 8 or NIHSS score of 0-2 in 24 (-2/+12) hours
Change in final cerebral infarct volume relative to baseline at 24 (-2/+12) hours postoperatively on CT/MR | 24 hours after thrombectomy
  Change in final cerebral infarct volume relative to baseline at 24 (-2/+12) hours postoperatively on CT/MR
Vascular recanalization | Immediately after thrombectomy
  Revascularisation assessed by DSA immediately after thrombectomy；Postoperative revascularisation assessed by CTA/MRA/DSA using Arterial Occlusive Lesion (AOL) grading at 24 (-2/+12) hours postoperatively；Application of bedside TCD for assessment of revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wei, doctorate, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China